CLINICAL TRIAL: NCT06211322
Title: The ReMonit Gout Feasibility Study
Brief Title: The Remote Monitoring of Gout Feasibility Study
Acronym: ReMonit Gout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Nina Osteras, Professor, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23/02662; 2023054 (Other Grant/Funding Number: South-Eastern Norway Health Authority)
Record Dates: First submitted 2023-12-20; First posted 2024-01-18 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- To determine the feasibility of a patient self-management application (Urika) in patients with gout. (Experimental): The intended purpose of the app is to support self-management for patients with gout that initiate urate lowering therapy.
  Interventions: Device: "Urika", a self-management application for patients with gout

INTERVENTIONS:
Device: "Urika", a self-management application for patients with gout — The self-management software application (Urika) will include information videos on gout and treatment, reminders of daily medication and blood tests, a built-in algorithm for medical dosage escalation, visualization and log of serum urate levels, motivational gamification, asynchronous chat function patient-health professionals, and a platform for remote monitoring by health professionals.

SUMMARY:
In this feasibility trial, a digital follow-up treatment strategy with patient self-management app (Urika) and remote monitoring in specialist healthcare for patients with gout will be tested.

DETAILED DESCRIPTION:
In this feasibility study various outcome measures will be assessed to determine whether the app (Urika) is viable, practical, and useful. The study will include assessments of technical, operational, clinical, and trial aspects of feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female >18 years of age at screening
* Patients with a clinical diagnosis of gout
* Patients who fulfil the American College of Rheumatology (ACR)/EULAR classification criteria
* Serum urate level >360 μmol/L at inclusion
* Having a smartphone/tablet

Exclusion Criteria:

* Contraindication for urate lowering therapy
* Unstable medical conditions (e.g,, uncontrollable hypertension, impaired liver function); known stage 3b or higher chronic kidney disease (estimated glomerular filtration (eGFR) rate/creatinine clearance <45 mL/min); severe infection or gastrointestinal bleed
* Major co-morbidities (e.g., malignancies, severe cardiovascular disease, severe diabetes mellitus, severe respiratory diseases)
* Psychiatric or mental disorders, alcohol abuse or other substance abuse, language barriers or other factors which makes adherence to the study protocol difficult

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Desirable feasibility level | Through study completion, an average of 3 months
  Acceptable overall feasibility of the app with ≥70% of the secondary endpoints indicating feasibility.

SECONDARY OUTCOMES:
App performance and functionality | Through study completion, an average of 3 months
  Acceptable number of errors (≤5 errors per participant) in the performance and functionality experienced by the patients and project group members
Patient-reported software usability | At 3 months
  Considered feasible if the System Usability Scale median score is ≥68 on a 0-100 scale, 100= best score
Patient-reported experiences and perceived benefits with the app | At 3 months
  Open responses will be collected in semi-structured interview. No scales or instruments will be used
Patient and health professionals' training requirements | Pre-baseline for health professionals and at baseline for patients
  Measured by registering amount of time spent (minutes) on training
Patient-reported satisfaction with the app | At 3 months
  Measured by a numeric rating scale (NRS) 0-10, higher scores mean better outcome. Acceptable feasibility if >=70% of the participants report score >=5, otherwise considered not acceptable feasibility.
Integration of workflow for health professionals | At screening and enrollment
  Measured by registering time spent on screening and enrollment
Serum urate level | At 3 months
  Considered feasible if there is available data on serum urate levels for ≥90% of patients for calculation of mean levels and proportion with low serum urate level
Patient-reported software functionality | Through study completion, an average of 3 months
  Total number of reported errors related to the software functionality (e.g., downloading, login, registration of medication, reminders, access to videos, medication adherence, registration of blood test results, urate level graph, blood test history, chat, request new prescription). Considered acceptable feasibility if the number of errors are ≤5 per patient in the performance and functionality experienced by the patients and project group members.
Urate lowering therapy dose escalation | Through study completion, an average of 3 months
  Considered feasible if patient-reported data and the medication history in the app monitored in the platform for health personnel is available for ≥90% of patients.
Patient-reported adherence to serum urate lowering therapy | At 3 months
  Patient-reported Medication Adherence Report Scale (MARS-5), score range 5-25, higher scores mean better adherence. Considered acceptable feasibility if >=90% of the patients complete the instrument.
Acute gout flares | At 3 months
  Number of acute gout flares
Side-effects of urate lowering therapy | At 3 months
  Number of side-effects registered in the app or by study nurse or study coordinator
Adverse events | At 3 months
  Number of adverse events (incl. serious adverse events) registered by study medical doctor, study nurse or study coordinator
Patient satisfaction with the follow-up care | At 3 months
  Measured by a single item with 5 response categories, ranging from very dissatisfied to very satisfied, higher scores mean higher satisfaction. Considered acceptable feasibility if >=70% of the participants report to be satisfied or very satisfied.
Knowledge of gout and recommended treatment | At baseline and 3 months
  Measured by the Gout Knowledge Questionnaire, 0-10, higher scores mean better outcome. Considered acceptable feasibility if there is available total score data for >=90% of the patients.
Pain related to gout | At 3 months
  Measured by a numeric rating scale (NRS) 0-10, lower scores mean better outcome. Considered acceptable feasibility if there is available data for >=90% of the participants.
Health related quality of life | At 3 months
  Measured by the Euro Quality of Life 5 Dimensions 5 Levels, each item is scored 1-5, lower scores mean better outcome. Considered acceptable feasibility if there is available data for >=90% of the participants.
Activity limitations | At 3 months
  Measured by Work Productivity and Activity Impairment (WPAI) item no.6, 0-10, lower scores mean better outcome. Considered acceptable feasibility if there is available data for >=90% of the participants.
Number of consultations in specialist or primary healthcare | At 3 months
  Considered acceptable feasibility if there is available data for ≥90% of patients on patient-reported visits in specialist or primary healthcare
Costs and time for traveling | At 3 months
  Considered acceptable feasibility if there is available data for ≥90% of patients on patient-reported time for travelling to the hospital
Sick leave and time off work | At 3 months
  Considered acceptable feasibility if there is available data for ≥90% of participants using self-report
Eligible patients per month | At enrollment
  Number of eligible patients per month.
Recruitment rate | After enrollment
  Acceptable recruitment rate is ≥50% of eligible patients.
Patient dropout | At 3 months
  Number of patients that withdraw from the study. Acceptable withdrawal rate is ≤20% of included patients.
Trial logistics | At 3 months
  Acceptable overall trial logistics (Identification, screening, recruitment, patient training, data collections, monitoring blood test results, renewal of prescriptions) evaluated as Yes vs. No by the study group.
Patients' app use: videos watched | Through study completion, an average of 3 months
  Count the number of videos watched per participant. Considered acceptable feasibility if ≥70% of the participants have watched at least 1 video.
Patients' app use: registrations of daily medication adherence | Through study completion, an average of 3 months
  Count the number of registrations of daily medication adherence. Considered acceptable feasibility if ≥70% of the participants have registered at least 1 adherence.
Patients' app use: registration of serum urate levels | Through study completion, an average of 3 months
  Count the number of registered serum urate levels. Considered acceptable feasibility if ≥90% of the patients register their serum urate level monthly.
Patients' app use: chat messages | Through study completion, an average of 3 months
  Count the number of chat messages. Considered acceptable feasibility if ≥70% of the participants register at least 1 chat message.
Patients' app use: flare registering | Through study completion, an average of 3 months
  Count the number of flare registering. Considered acceptable feasibility if ≥10% of the participants register 1 flare.
Potential risk and challenges | At 3 months
  Incidence of hinders that could harm a successful clinical evaluation of the app in a large randomised, controlled trial.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Østerås, Prof., Principal Investigator — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway